CLINICAL TRIAL: NCT00752102
Title: A Phase IV, Randomized, Single-center Study of the Effects of Calcitriol and Paricalcitol on Vascular Calcification in Chronic Kidney Disease Stages 3 and 4
Brief Title: Vitamin D and Coronary Calcification Study
Acronym: VCOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Abbott #20128
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Chronic Kidney Disease; Vitamin D Deficiency; Coronary Calcification; Disorders of Calcium and Bone Metabolism
Keywords: Secondary Hyperparathryoidism; Chronic Kidney Disease; Vitamin D; Coronary Calcification; Bone metabolism
MeSH Terms: conditions — Renal Insufficiency, Chronic; Vitamin D Deficiency | interventions — Calcitriol; paricalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcitriol (Active Comparator): Calcitriol is a synthetic vitamin D analog which is active in the regulation of the absorption of calcium from the gastrointestinal tract and its utilization in the body. Calcitriol is available as capsules containing 0.25 mcg or 0.5 mcg calcitriol and as an oral solution containing 1 mcg/ml of calcitriol. All dosage forms contain butylated hydroxyanisole (BHA) and butylated hydroxytoluene (BHT) as antioxidants.
  Subjects taking calcitriol started at 0.25 mcg 3x/week and titrated up during the next visit according to PTH levels.
  Interventions: Drug: Calcitriol (Rocaltrol®)
- Paricalcitol (Active Comparator): Paricalcitol, USP, the active ingredient in Zemplar® Capsules, is a synthetically manufactured analog of calcitriol, the metabolically active form of vitamin D indicated for the prevention and treatment of secondary hyperparathyroidism in chronic kidney disease. Zemplar is available as soft gelatin capsules for oral administration containing 1 mcg, 2 mcg or 4 mcg of paricalcitol. Each capsule also contains medium chain triglycerides, alcohol, and butylated hydroxytoluene.
  Subjects taking paricalcitol will be started at 2 mcg 3x/week and titrated up during the next visit according to PTH levels.
  Interventions: Drug: Paricalcitol

INTERVENTIONS:
Drug: Calcitriol (Rocaltrol®) — Subjects taking calcitriol will be started at 0.25 mcg 3x/week and titrated up during the next visit according to PTH levels. If at the 12 week visit, PTH is still not at goal, then calcitriol will be increased to 0.5 mcg 3x/week.
  Other Names: Calcijex®; Rocaltrol®
  Arms: Calcitriol
Drug: Paricalcitol — Subjects taking paricalcitol will be started at 2 mcg 3x/week and titrated up during the next visit according to PTH levels. If at the 12 week visit, PTH is still not at goal, then paricalcitol will be increased to 4 mcg 3x/week.
  Other Names: Zemplar®
  Arms: Paricalcitol

SUMMARY:
Patients with chronic kidney disease (CKD) have a higher mortality rate than the general population, with cardiovascular disease (CVD) accounting for approximately 50% of deaths. Vascular calcification is a common finding in patients with CKD. Furthermore, patients with CKD develop secondary hyperparathyroidism, partly because of a decrease of calcitriol synthesis on the kidney. Treatment of secondary hyperparathyroidism includes use of activated vitamin D including calcitriol and paricalcitol. Recent evidence in dialysis patients suggest an improved survival in patients using paricalcitol compared to calcitriol.

Studies in uremic rats suggests that there are differential effects of calcitriol and paricalcitol in expression of markers of soft-tissue calcification independent of calcium-phosphorus product. Calcitriol increased calcification of vascular smooth muscle cells cultured in calcification media. There was also significant increase in pulse pressure in animals treated with calcitriol.

The investigators hypothesize that these different forms of vitamin D may have differential effects in vascular calcification progression in CKD patients.

DETAILED DESCRIPTION:
Coronary artery calcification (CAC) is a risk marker for CVD and mortality. In animal models, calcitriol significantly increased the serum calcium-phosphate product and aortic calcium content, while paricalcitol had no effect. The objective of this randomized, blinded single-center is to determine the differential effect of oral calcitriol and paracalcitol on vascular calcification in patients with chronic kidney disease (CKD).

We performed a total of 89 screening visits and randomized 44 participants. Forty participants completed the final visit. Diagram 1 presents the recruitment schematic.

ELIGIBILITY:
Inclusion Criteria:

* CKD stages 3 or 4 (estimated glomerular filtration rate (eGFR) between 15 and 59)
* Diagnosis of secondary hyperparathyroidism, which is defined as:

  * Elevated intact PTH (iPTH) as per KDIGO guidelines:

    * CKD stage 3 (eGFR 30-59) or CKD stage 4 (eGFR 15-29) with iPTH > Upper Limit of Normal for lab (6.8 pmol/L)
* Presence of Coronary Artery Calcium (CAC > 0)
* Subject will be able to complete the study, to the best of his/her knowledge

Exclusion Criteria:

* iPTH >1500 pg/ml
* Current or previous use of bisphosphonates
* History of parathyroidectomy or anticipated parathyroidectomy
* History of cinacalcet use
* History of a solid organ transplant or scheduled date for transplant surgery
* History of coronary revascularization (coronary artery bypass surgery or percutaneous intervention)
* History of coronary artifact (e.g. pacemaker, intracardiac defibrillator, artificial valve or biventricular leads)
* Active atrial fibrillation
* Weight greater than 300 pounds (due to limitations of equipment)
* HIV positive
* Current pregnancy (although pregnancy is very rare in the CKD population)
* Life expectancy less than two years as judged by primary physician
* Institutionalized patients (nursing home or prisoners)
* Language barrier or mental incapacity to consent
* Inability to swallow tablets or current gastrointestinal disorder that may be associated with impaired absorption of orally administered medications.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia E Rosas, MD, MSCE, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Anis KH, Pober D, Rosas SE. Vitamin D Analogues and Coronary Calcification in CKD Stages 3 and 4: A Randomized Controlled Trial of Calcitriol Versus Paricalcitol. Kidney Med. 2020 Jun 17;2(4):450-458. doi: 10.1016/j.xkme.2020.05.009. eCollection 2020 Jul-Aug. PMID 32775985

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calcitriol | Paricalcitol
Started | 22 | 22
Completed | 19 | 21
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcitriol | Paricalcitol | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 65.8 (7.4) | 65.5 (11) | 65.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 18
  Male | 17 | 9 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 15 | 29
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Coronary Artery (CAC) Score Progression
Description: coronary artery (CAC) score difference between baseline and followup CT scans. It was measured in Agatston units. These are units of amount of calcification in the blood vessels so it's a continuous variable. The amount of calcium was quantified with the Agatston scoring method. Calcium scores were adjusted with a standard calcium phantom that was scanned along with the participant. The phantom contained known calcium density bars and provided a way to calibrate the x-ray attenuation level.
  Participants scoring CAC >400 are considered to be at risk for having at least one coronary lesion.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: Agatston units
Arm/Group | Calcitriol | Paricalcitol
Number analyzed (Participants) | 19 | 21
Agatston units | 74.38 (110.39) | 106.32 (126.06)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the time between scans (0-48 weeks)
Arm/Group | Calcitriol | Paricalcitol
All-Cause Mortality (participants affected / at risk) | 2/22 | 1/22
Serious Adverse Events (participants affected / at risk) | 9/22 | 8/22
Other Adverse Events (participants affected / at risk) | 18/22 | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcitriol (N=22) | Paricalcitol (N=22)
hospitalization for congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Dialysis Initiation (Renal and urinary disorders) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 1 (1) | 0 (0)
Hypotensive Episode (Cardiac disorders) | 1 (1) | 0 (0)
Prostatectomy and Laparoscopic Lymph node Dissection (Surgical and medical procedures) | 1 (1) | 0 (0)
Lower Urinary Tract Symptoms, bladder mass. low grade urothelial carcinoma of bladder, cystoscopy (Renal and urinary disorders) | 1 (1) | 0 (0)
Hip dislocation (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Hip Replacement Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Psychiatric Hospitalizaton (Psychiatric disorders) | 1 (1) | 0 (0)
Broken Patella in trip and fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Prostate Cancer (Renal and urinary disorders) | 1 (1) | 0 (0)
Chest pain due to cocaine use, Congestive Heart Failure and Shortness of breath (Cardiac disorders) | 0 (0) | 1 (2)
Congestive Heart Failure Exacerbation (Cardiac disorders) | 0 (0) | 1 (1)
Hemodialysis access surgery (Renal and urinary disorders) | 0 (0) | 2 (2)
Hypercapnic/hypercarbic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypercarbic respiratory failure - diastolic dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ER visit for new CPAP mask (Surgical and medical procedures) | 0 (0) | 1 (1)
Asthma Exascerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ER visit: fall at home causing back and flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Hypercarbic respiratory failure, pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hospitalization - gastroesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
TIA, confusion (Nervous system disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Gout flare (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia; acute on chronic kideney failure (Renal and urinary disorders) | 0 (0) | 1 (1)
ED visit - 2nd right toe infection (Infections and infestations) | 0 (0) | 1 (1)
Hypoglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Started hemodialysis (Renal and urinary disorders) | 0 (0) | 1 (1)
Uncontrolled blood pressure atime of study - took her to ER (Cardiac disorders) | 0 (0) | 1 (1)
ER Visit - Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcitriol (N=22) | Paricalcitol (N=22)
Viral Upper Respiratory Illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fatigue (Nervous system disorders) | 1 (1) | 3 (3)
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hip Dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fistula Placement (Renal and urinary disorders) | 1 (1) | 0 (0)
Broken Patella in trip and fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute Fever s/p biopsy (General disorders) | 1 (1) | 0 (0)
Visicoli placement surgery for prostate cancer treatment (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hand and leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mild hyperkalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Spontaneous right conjunctival bleed (Eye disorders) | 1 (1) | 0 (0)
Forgetful, "something wrong with head" (Nervous system disorders) | 1 (1) | 0 (0)
Left eye cataract extraction (Eye disorders) | 1 (1) | 0 (0)
Nocturnal Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Right eye cataract extension (Eye disorders) | 1 (1) | 0 (0)
Left Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
2 episodes chest pain while lying down for bed (Cardiac disorders) | 1 (1) | 0 (0)
hyperphosphatemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Shortness of Breath, Fatigue (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elevated BP and Edema (Cardiac disorders) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea & vomiting, fatigued, shortness of breath (Gastrointestinal disorders) | 1 (1) | 1 (1)
Blunt head injury, hip pain following fall from chair (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in left leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Edema & generalized pain left foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ankle sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperkalemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Uremia Symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Headaches, fatigue (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 4 (9)
Gout flare (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Weakness, fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cataract Surgery (Eye disorders) | 1 (1) | 0 (0)
Loose stool in AM (Gastrointestinal disorders) | 1 (1) | 0 (0)
Metal taste (Gastrointestinal disorders) | 2 (2) | 3 (6)
Kidney pain/ kidney stones (Renal and urinary disorders) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (2) | 0 (0)
ER visit (depression exacerbation) (Psychiatric disorders) | 1 (1) | 0 (0)
Swollen Elbow (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Diffuse low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest pain, possible muscle pull (Cardiac disorders) | 0 (0) | 1 (1)
Edema (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Uremic symptoms (Renal and urinary disorders) | 0 (0) | 1 (1)
AVF placement (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 3 (3)
Night Sweats (Nervous system disorders) | 0 (0) | 1 (1)
Increased thirst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hospitalization with UTI (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Replacement of nephrostomy tube (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Increased Edema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dizzy, diadiaphoretic, fall in anemia clinic (Nervous system disorders) | 0 (0) | 1 (1)
Severe gout in left foot (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Azotemia, hyperkalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Back pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anorexia in AM (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Persistent edema (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Nausea, vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypercalcemia (Endocrine disorders) | 0 (0) | 1 (1)
Hyperphosphatemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Poison ivy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cataract extraction & lens implantation (Eye disorders) | 0 (0) | 1 (1)
knee pain due to fall on bus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Indeterminate left renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Nausea & fatigue on passing a stone (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Worsening flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Broken right foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Feels faint in morning (Nervous system disorders) | 0 (0) | 1 (1)
ED Visit - CHF, foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
gout flare (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Problems going to the bathroom (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Little headache with unbalance (Nervous system disorders) | 0 (0) | 1 (1)
Tingling in arms (Nervous system disorders) | 0 (0) | 1 (1)
Fleeting dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Fistula placement (Renal and urinary disorders) | 0 (0) | 1 (1)
Fall at phleobtomy suites (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LE cellulitis (Infections and infestations) | 0 (0) | 1 (1)
TDC Cath placement (Renal and urinary disorders) | 0 (0) | 1 (1)
Long QT (Cardiac disorders) | 0 (0) | 1 (1)
Arthritis pain left knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leg cramping and pains (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Broken toe (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hematoma on knee (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bronchitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No